CLINICAL TRIAL: NCT02769234
Title: ERP and qEEG Measures Collected in Outpatient Settings as Indices of Disease Progression in Alzheimer's Disease (AD)
Brief Title: EEG/ERP Longitudinal Study in Alzheimer's Disease (AD)
Status: Completed | Type: Observational
Sponsor: Neuronetrix, Inc. (Industry)
Collaborators: Boston Center for Memory (Unknown); The Memory Clinic of Vermont (Unknown); Premiere Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: SRP-1782
Record Dates: First submitted 2015-02-26; First posted 2016-05-11 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Alzheimer's Disease
Keywords: EEG; ERP; Event-related Potentials; Alzheimer's; P300
MeSH Terms: conditions — Alzheimer Disease | interventions — Psychometrics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alzheimer's disease: Subjects with a diagnosis of Alzheimer's disease that successfully performed an ERP/EEG test with the COGNISION(TM) System prior to enrollment for the current study are eligible to participate.
  Interventions: Procedure: ERP/EEG test; Procedure: Psychometric testing

INTERVENTIONS:
Procedure: ERP/EEG test — The testing protocol consists of an auditory oddball ERP paradigm, followed by the collection of 3min of resting EEG. During the ERP paradigm a variety of auditory stimuli are played through the system's earphones while voltage potentials are recorded from the subject's scalp. At the end of the ERP session, 3 minutes of EEG data will be recorded while the subject is resting. The entire procedure, including set up, instructions to the subject and actual test is expected to take 45-60 minutes.
Procedure: Psychometric testing — Subjects that complete ERP/qEEG testing successfully will move on to clinical and neuropsychological evaluation. Demographic information with also be collected.

SUMMARY:
In a previous study, NCT00582127, two age-matched cohorts, one clinically diagnosed with mild Alzheimer's disease and the other healthy controls, were tested with a hand-held EEG/ERP system to determine if the cohorts could be discriminated using the EEG/ERP measures. This study proposes to retest the AD cohort 18-60 months after their first test to characterize the change in EEG/ERP measures correlated with the longitudinal change in neuropsychological testing.

DETAILED DESCRIPTION:
In study NCT00582127, two age-matched cohorts (mild AD, n=98 and healthy controls, n=100) were recruited to 7 clinical sites to undergo a broad range of clinical, neuropsychological, and neuroelectrophysiological tests. The complete battery of ADNI neuropsychological tests were performed on the mild AD subjects as well as standard blood tests and MRI using the ADNI protocol. MRI volumetry analysis was performed on the MRI data. Both cohorts underwent a 3-minute EEG recording and event-related potential (ERP) testing using a standard 2-deviant auditory oddball paradigm with the COGNISION(tm) System from Neuronetrix. The study showed that specific EEG/ERP features could be used to discriminate the mild AD cohort from healthy controls.

The current study is intended as a follow up to NCT00582127.AD subjects that successfully completed COGNISION™ and psychometric testing in the previous study are eligible to be part of the present follow up.

In the first part of the current study, de-identified cognitive and functional data for the AD patients that the sites have collected during regular check ups after testing for the original Neuronetrix study will be shared with the study Sponsor. The retrospective chart review has three main objectives:

* Quantify the rate of cognitive and functional decline in these patients.
* Investigate whether ERP and/or qEEG data collected during testing for the original Neuronetrix study can provide any insight on subsequent rate of cognitive and functional decline.
* Identify study subjects that might still be functional enough to successfully complete a follow-up ERP/qEEG test. These subjects will be offered an opportunity to come back to the sites for follow-up ERP/qEEG and psychometric testing.

Up to 40 subjects will be invited back to the sites. Subjects that choose to enroll in the second part of the study will have an ERP/qEEG test administered by a Neuronetrix certified test administrator. Subjects that complete the test successfully will move on to clinical evaluation and psychometric testing.

Results obtained from this part of the study will be compared with ERP/qEEG and psychometric data from the completed Neuronetrix study mentioned above. The two main objectives of the comparisons will be:

* Investigate whether ERP and qEEG measures collected in outpatient settings show significant changes over time in subjects with AD.
* Correlate longitudinal changes in ERP and qEEG measures (if any) with cognitive and functional decline as measured by psychometric tests.

ELIGIBILITY:
Inclusion criteria:

Between 60 and 95 years old (inclusive) A diagnosis of Alzheimer's disease A successful ERP/EEG test performed with the COGNISION™ system 2-5 years prior to testing for the current study

A sub-group of up to 40 subjects will be called back to the sites for follow-up ERP/qEEG and psychometric testing. Additional inclusion criteria for these subjects will be:

* Willing and able to undergo ERP/EEG and psychometric testing
* Have a study partner able to provide an independent evaluation of functioning
* Permitted medications stable for at least 2 weeks prior to testing

Exclusion Criteria:

Subjects will not be called back to sites for follow-up testing if they have:

* Known allergy to latex
* Neuropsychological tests administered within three months of study enrollment
* Investigational agents administered within three months of study enrollment
* Severe cognitive and functional deficits that in the judgement of the site PI will prevent them from successfully completing ERP/EEG and/or psychometric testing
* Any significant systemic illness or unstable medical condition at the time of testing which could lead to difficulty complying with the protocol
* Use of psychoactive substances (Gingko Biloba, melatonin, sedatives etc.) will be allowed as long as the subject suspends their use on the day of testing. Smokers will not be required to abstain.

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AD subjects that successfully completed ERP/EEG testing during NCT00582127.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-05; Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Correlation (longitudinal change) between EEG/ERP vs. Neuropsychological Testing. | 24-60 Months

SECONDARY OUTCOMES:
Correlation (longitudinal change) between EEG/ERP vs ADNI-EF composite. | 24-60 Months
Correlation (longitudinal change) between EEG/ERP vs. ADNI-Mem composite. | 24-60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Marco Cecchi, PhD, Study Director — Neuronetrix, Inc.
Locations (3):
- United States (3):
  - Premiere Research Institute, West Palm Beach, Florida
  - Boston Center for Memory, Brookline, Massachusetts
  - The Memory Clinic, Bennington, Vermont

REFERENCES:
- [Background] Cecchi M, Moore DK, Sadowsky CH, Solomon PR, Doraiswamy PM, Smith CD, Jicha GA, Budson AE, Arnold SE, Fadem KC. A clinical trial to validate event-related potential markers of Alzheimer's disease in outpatient settings. Alzheimers Dement (Amst). 2015 Oct 2;1(4):387-94. doi: 10.1016/j.dadm.2015.08.004. eCollection 2015 Dec. PMID 27239520